CLINICAL TRIAL: NCT06149260
Title: An Open-lable Trial of Subcutaneous Semaglutide in Systemic Scleroderma
Brief Title: Subcutaneous Semaglutide in Systemic Scleroderma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Rong Xiao, Professor of Dermatology, MD, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYG2022061
Record Dates: First submitted 2023-11-16; First posted 2023-11-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Scleroderma, Systemic; Fibrosis; Semaglutide
MeSH Terms: conditions — Scleroderma, Systemic; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Semaglutide (Experimental): Participants will receive once-weekly semaglutide subcutaneous injection at escalating doses from 0.25 mg/week to 0.5 mg/week.
  Interventions: Drug: Semaglutide Pen Injector

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Inject semaglutide subcutaneously once weekly, on the same day each week, at any time of day, in a dose increasing mode: the initial dose of 0.25mg QW (once a week), increased to 0.5mg QW after 4 weeks, and then maintained 0.5mg until the end of treatment in total 24 weeks.

SUMMARY:
This trial will study the safety and efficacy of subcutaneous semaglutide for the treatment of Systemic Sclerosis

DETAILED DESCRIPTION:
Systemic Sclerosis (Ssc) is a rare, systemic autoimmune disease characterized by skin fibrosis and vasculopathy. In addition to the skin, it is a heterogeneous disease that affects multiple organs, including the cardiac, pulmonary, and gastrointestinal systems. This is a small prospective and open-label clinical trial of semaglutide in adults with systemic slceorsis. 10 systemic sclerosis patients will be recruited and receive semaglutide for 24 weeks. The primary endpoint of the study is the change in mRSS at 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:(Those who have not achieved good results after hormone or immunosuppressive therapy)

1. Gender unlimited;
2. Age 18-65 years old (including 65 years old);
3. Patients diagnosed with SSc who meet the 2013 European Union Against Rheumatology (EULAR)/American Society of Rheumatology (ACR) SSc diagnostic classification criteria and exclude infections, tumors, and other connective tissue diseases.
4. Has received one or more of the following standard systemic treatments allowed by the research protocol:

   1. Before the first subcutaneous injection of the study, oral corticosteroids (prednisone not exceeding 15mg/d or equivalent) were administered for ≥ 8 weeks, and stabilizers were administered for ≥ 4 weeks.
   2. Before the first subcutaneous injection of the study, patients were treated with Tofacitinib (5-10mg/d) for ≥ 8 weeks and received a stabilizer dose for ≥ 6 weeks.
   3. If one or more of the following immune modulators are used, treatment must be given for ≥ 12 weeks before the start of the study, and treatment with a stabilizer dose must be given for ≥ 6 weeks Oral mycophenolate mofetil (MMF) ≤ 1.5 g/day Methotrexate (MTX) oral ≤ 15 mg/week, combined with folic acid Cyclosporine If the subjects use ≥ 2 of the above immunomodulatory drugs in combination, the appropriateness of the subjects' participation in the study must be discussed with the medical supervisor and study chair before enrollment.
5. A modified Rodnan Skin Score (mRSS) of > 14
6. Those who sign an informed consent form, voluntarily participate in this project, and are able to complete follow-up as required.

Exclusion Criteria:

1. Prior to the first dose, Body Mass Index (BMI) < 18.5 kg/m2; weight loss of 10% within one month or 20% within six months.
2. Family or personal history of type 2 multiple endocrine neoplasia or medullary thyroid carcinoma, with family history involving first-degree relatives.
3. History of malignant tumors or a history of malignant tumors within the past 5 years before screening.
4. Presence of other inflammatory diseases that may interfere with efficacy assessment, including but not limited to rheumatoid arthritis (RA), overlap syndrome, psoriasis, dermatomyositis, multiple sclerosis, Crohn's disease, or active Lyme disease.
5. Severe gastrointestinal complications of systemic sclerosis (SSc), such as significant swallowing difficulties, and severe diseases affecting vital organ systems such as the heart, brain, lungs, liver, kidneys, or blood, as deemed unsuitable for participation in the study by the investigator.
6. Known current active or recurrent severe infections, including active tuberculosis.
7. Congenital immunodeficiency or congenital immunosuppression.
8. Substance abuse, alcoholism, or psychiatric disorders, rendering patients uncooperative or unable to adhere to treatment; poor predictability of compliance.
9. Women who are pregnant, breastfeeding, or planning to become pregnant.
10. Patients currently participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-08-29 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in modified Rodnan skin score (mRSS) at week 24 | Baseline and 24 weeks
  Change in modified Rodnan skin score (mRSS) at week 24 performed by the same investigator at week 0 and week 24 and the change in mRSS will be calculated following the formula: ΔmRSS= mRSSw24 - mRSSw0.
  To measure mRSS, skin thickness of the patient is rated by palpation at each of 17 anatomic sites using a scale of 0-3 (0 = normal skin; 1= mild thickness; 2= moderate thickness; 3=severe thickness with an inability to pinch the skin into a fold). The scores at each site are summed with a minimum of 0 and a maximum of 51 (17 sites)

SECONDARY OUTCOMES:
Incidence of Adverse Events | Baseline and 24 weeks
Incidence of Severe Adverse Events | Baseline and 24 weeks
the scleroderma health assessment questionnaire-disability index (sHAQ-DI) | Baseline and 24 weeks
High-resolution computer tomography (HRCT) | Baseline and 24 weeks
Forced Vital Capacity(FVC) and Diffusing capacity of the lung for carbon monoxid(DLCO) | Baseline and 24 weeks
St George' s Respiratory Questionnaire(SGRQ) | Baseline and 24 weeks
Pulmonary arterial hypertension by echocardiography | Baseline and 24 weeks
left ventricular ejection fraction by echocardiography | Baseline and 24 weeks
6-Minute Walk Test (6MWT) Distance | Baseline and 24 weeks
gastrointestinal tract (GIT) in scleroderma score | Baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rong Xiao, MD, Study Chair — Department of Dermatology, Second Xiangya Hospital of Central South University, Changsha, China; Licong Liu, MD, Principal Investigator — Second Xiangya Hospital; Yaqian Shi, MD, Principal Investigator — Second Xiangya Hospital; Zhuotong Zeng, MD, Principal Investigator — Second Xiangya Hospital; Zhan Yi, MD, Principal Investigator — Second Xiangya Hospital; Xiangning Qiu, MD, Principal Investigator — Second Xiangya Hospital; Ruixuan Zhu, MD, Principal Investigator — Second Xiangya Hospital; Yi Wei, MD, Principal Investigator — Second Xiangya Hospital; Ke Chai, MD, Principal Investigator — Second Xiangya Hospital; Hao Ren, MD, Principal Investigator — Second Xiangya Hospital; Yangfan Xiao, MD, Principal Investigator — Second Xiangya Hospital
Locations (1):
- the Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No